CLINICAL TRIAL: NCT03858192
Title: Understanding Acute Sarcopenia: a Time-limited Cohort Study to Characterise Changes in Muscle Mass and Physical Function in Older Adults Following Hospitalisation
Brief Title: Understanding Acute Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Dowager Countess Eleanor Peel Trust (Unknown); University Hospital Birmingham NHS Foundation Trust (Other); MRC-Arthritis Research UK Centre for Musculoskeletal Ageing Research (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RG_18-213
Record Dates: First submitted 2019-02-08; First posted 2019-02-28 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-01

CONDITIONS: Sarcopenia
Keywords: Acute sarcopenia, muscle, physical function, older adults
MeSH Terms: conditions — Sarcopenia | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elective colorectal surgery (Experimental): Patients who are expected to undergo a major colorectal surgery procedure will be recruited to this study preoperatively and followed-up until three months postoperatively.
  Interventions: Procedure: Colorectal surgery procedure
- Emergency abdominal surgery (Experimental): Patients who are admitted as an emergency and undergo abdominal surgery will be recruited from general surgery wards either preoperatively or within 48 hours of surgery. They will be followed-up until three month postoperatively.
  Interventions: Procedure: Emergency abdominal surgery
- Medical patients (Experimental): Patients admitted under general medicine with an infection will be recruited from general medicine wards within 48 hours of admission. They will be followed-up until three month post-admission
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Procedure: Colorectal surgery procedure — Elective admission for colorectal surgery
  Arms: Elective colorectal surgery
Procedure: Emergency abdominal surgery — Emergency admission necessitating emergency surgery
  Arms: Emergency abdominal surgery
Drug: Antibiotics — Treatment for infection and reason for admission
  Arms: Medical patients

SUMMARY:
This study aims to characterise acute changes in muscle mass, strength, physical performance in hospitalised older adults. We will assess the impact of these changes upon physical function at three month follow-up, and assess for the impact of clinical and immune-endocrine factors upon these changes.

DETAILED DESCRIPTION:
Study Design

Time-limited cohort study involving serial measurements of Bilateral Anterior Thigh Thickness (BATT) using ultrasound, handgrip strength, physical performance, and physical function measured using the Patient Reported Outcome Measures Information System (PROMIS®). We aim to fully characterise changes in these patients, and will perform a comprehensive evaluation of clinical factors including nutrition and physical activity, and measure immune-endocrine markers of inflammation.

Study Participants

Elective colorectal surgery, emergency abdominal surgery, and medical patients aged 70 years and older

Planned Size of recruitment target

56 elective colorectal patients, 56 emergency abdominal surgery patients, and 56 medical patients with acute infections

Follow up duration

3 months

Primary research question

Does acute change in quadriceps muscle thickness, handgrip strength and/or physical performance within one week of hospitalisation predict change in patient reported physical function at three months?

ELIGIBILITY:
Inclusion Criteria:

ELECTIVE COHORT

* Aged 70 years or older at time of recruitment
* Expected to undergo an elective major colorectal surgery procedure

EMERGENCY SURGERY COHORT

* Aged 70 years or older at time of recruitment
* Emergency admission
* Expected to undergo emergency abdominal procedure during admission, or emergency abdominal procedure performed within previous 48 hours

MEDICAL COHORT

* Aged 70 years or older at time of recruitment
* Emergency admission for acute bacterial infection or presumed acute bacterial infection

Exclusion Criteria:

ELECTIVE COHORT

* Unable to provide written informed consent at time of recruitment
* Unable to understand verbal English
* Life expectancy less than 30 days

EMERGENCY SURGERY COHORT

* Unable to provide written informed consent at time of recruitment and no consultee available
* Unable to understand verbal English
* Life expectancy less than 30 days

MEDICAL COHORT

* Unable to provide written informed consent at time of recruitment and no consultee available
* Unable to understand verbal English
* Life expectancy less than 30 days

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2019-05-03 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Physical function | Three months
  Change in physical function at three months as measured by the T score derived from the Patient Reported Outcome Measures Information System (PROMIS®) - Item Bank v. 2.0, Physical Function, Short Form 10b.
  This is a patient-reported outcome measure of physical function. Raw scores are collected out of a maximum of 50; minimum of 10. These are converted to T scores, which are used for analysis (mean 50, SD 10; range 13.8 - 61.3). Higher scores are representative of better physical function.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Three months
  Change in Short Physical Performance Battery (SPPB) score at (elective cohort)
Bilateral Anterior Thigh Thickness (BATT) | Three months
  Change in BATT (elective and emergency cohorts)
Handgrip strength | Three months
  Change in handgrip strength (elective and emergency cohorts)
Acute changes during hospitalisation - gait speed | One week
  Change in gait speed within one week of hospitalisation (elective and emergency cohorts)
Acute changes during hospitalisation - BATT | One week
  Change in BATT within one week of hospitalisation (elective and emergency cohorts)
Acute changes during hospitalisation - handgrip strength | One week
  Change in handgrip strength within one week of hospitalisation (elective and emergency cohorts)
Rectus femoris echogenicity (quantified using ImageJ software) | Immediately postoperatively, one week postoperatively, and at three months
  Change in rectus femoris echogenicity (elective and emergency cohorts)
BATT: subcutaneous tissue ratio (BATT-SCR) | Immediately postoperatively and one week postoperatively
  Change in BATT: subcutaneous tissue ratio (BATT-SCR) (elective and emergency cohorts)
Acute sarcopenia | One week postoperatively
  Incidence of acute sarcopenia (elective and emergency cohorts)
Physical activity - steps taken | One week
  Postoperative physical activity (steps taken) as measured by physical activity recorders (subset of elective and emergency cohorts)
Physical activity - steps taken | One month
  Postoperative physical activity (steps taken) as measured by physical activity recorders (subset of elective and emergency cohorts)
Physical activity - distance walked | One week
  Postoperative physical activity (distance walked) as measured by physical activity recorders (subset of elective and emergency cohorts)
Physical activity - distance walked | One month
  Postoperative physical activity (distance walked) as measured by physical activity recorders (subset of elective and emergency cohorts)
Sedentary time | One week
  Postoperative sedentary time as measured by physical activity recorders (subset of elective and emergency cohorts)
Sedentary time | One month
  Postoperative sedentary time as measured by physical activity recorders (subset of elective and emergency cohorts)
Acceptability (objective) - refusal | Three months
  Participant refusal rates (elective and emergency cohorts)
Acceptability (objective) - missing data | Three months
  Missing data (elective and emergency cohorts)
Acceptability (objective) - drop-outs | Three months
  Drop-out rates (elective and emergency cohorts)
Acceptability (patient-reported) | Three months
  Total derived acceptability score as measured by questionnaire upon study completion (elective and emergency cohorts)

CONTACTS AND LOCATIONS:
Overall Officials: Carly Welch, MBChB, Study Director — University of Birmingham; Thomas Jackson, MBChB, PhD, Principal Investigator — University of Birmingham
Locations (1):
- Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Welch C, K Hassan-Smith Z, A Greig C, M Lord J, A Jackson T. Acute Sarcopenia Secondary to Hospitalisation - An Emerging Condition Affecting Older Adults. Aging Dis. 2018 Feb 1;9(1):151-164. doi: 10.14336/AD.2017.0315. eCollection 2018 Feb. PMID 29392090
- [Background] Welch C, Greig CA, Hassan-Smith ZK, Pinkney TD, Lord JM, Jackson TA. A pilot observational study measuring acute sarcopenia in older colorectal surgery patients. BMC Res Notes. 2019 Jan 14;12(1):24. doi: 10.1186/s13104-019-4049-y. PMID 30642375
- [Derived] Welch C, Greig C, Masud T, Jackson TA. Muscle quantity and function measurements are acceptable to older adults during and post- hospitalisation: results of a questionnaire-based study. BMC Geriatr. 2021 Feb 25;21(1):141. doi: 10.1186/s12877-021-02091-3. PMID 33632138
- [Derived] Welch C, Greig CA, Masud T, Pinkney T, Jackson TA. Protocol for understanding acute sarcopenia: a cohort study to characterise changes in muscle quantity and physical function in older adults following hospitalisation. BMC Geriatr. 2020 Jul 10;20(1):239. doi: 10.1186/s12877-020-01626-4. PMID 32650734
- See also: Overall project website (to be updated throughout course of study) — http://acutesarcopenia.wordpress.com